CLINICAL TRIAL: NCT02330146
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of RCT-01 in Men and Women With Unilateral, Chronic Achilles Tendinosis
Brief Title: Safety and Efficacy of RCT-01 in Men and Women With Unilateral, Chronic Achilles Tendinosis
Acronym: ReaCT
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: * slower than anticipated rate of enrollment
  * need to obtain safety and efficacy data in a timely manner
  * pending expiry of manufacturing materials/reagents
Sponsor: RepliCel Life Sciences, Inc. (Industry)
Collaborators: Syreon Corporation (Industry); Innovacell Biotechnologie AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RCT-01-001-2014
Record Dates: First submitted 2014-12-12; First posted 2015-01-01 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Tendinosis; Tendinopathy
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RCT-01 (Experimental): Cultured, autologous hair follicle cells suspended in cryomedium
  Interventions: Drug: RCT-01
- Placebo (Placebo Comparator): cryomedium
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RCT-01
  Arms: RCT-01
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to assess the safety profile of RCT-01 injections as compared to placebo injections. This study will also measure the impact these injections will have on tendon structure and function and the symptoms of Achilles tendinosis.

28 participants will be selected for this study based on their health status, current/past medications, and ability to adhere to protocol-related requirements. Prior to entering the screening phase of the study, all potential study participants will have had to have at least 3 months of therapy for their unilateral, chronic (symptoms >6 months) Achilles tendinosis directed by a certified physiotherapist without a clinical response. At the first visit and after providing informed consent participants are evaluated against the study inclusion/exclusion criteria and provide blood samples for screening assessments (including virology). If suitable for study participation, participants will provide a biopsy from the scalp from which RCT-01 will be prepared.

Baseline evaluations of participants' overall health and tendinosis, in particular, will be performed on the day of injection. Once all baseline assessments have been completed, the tendon to be treated will be anesthetized and will receive ultrasound-guided injections of either placebo (cryomedium) or RCT-01.

All participants will return to the clinic for repeat assessments of their unilateral Achilles tendinosis and overall health at seven (7) visits over the following 6 months. Participants will also complete an eccentric training physiotherapy program under the guidance of a certified physiotherapist for two (2) months after receipt of injections. Total duration of patient participation is approximately eight (8) months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the age of 18 and 65 years and in good health having evidence of mid-substance unilateral, chronic Achilles tendinosis confirmed by ultrasound imaging.
2. Participant confirmation of symptoms of unilateral chronic Achilles tendinosis for at least 6 months
3. Completion of at least three months of physiotherapy for treatment of Achilles tendinosis at the study tendon as directed by a certified physiotherapist.
4. VISA-A score of less than 70 at Visit S1.
5. Willingness to provide written informed consent for participation in the study, attend all study visits and complete all procedures required by this protocol.
6. Fluent understanding of written and spoken English language
7. Females must either be post-menopausal for at least one year, surgically sterile, or, if of childbearing potential, using highly-effective methods of birth control during the study. This method of contraception must be used at least 4 weeks prior to screening (Visit S1) and during the entire duration of the clinical trial.

Exclusion Criteria:

1. Any prior therapeutic injections to the Achilles tendon to be studied (e.g., platelet-rich plasma, prolotherapy, dextrose, dry needling, etc) within 6 months of study Visit S1.
2. History of Achilles tendon surgery (either tendon)
3. Presence of enthesopathy or insertional tendinopathy in any tendons of the lower extremity, including Achilles tendons.
4. Presence of any medical condition that influences lower extremity function (e.g. osteoarthritis, presence of any peripheral nerve involvement, etc.)
5. Presence of seronegative arthropathies, diabetes mellitus (type I and II), elevated blood sugar, insertional arthropathies-psoriasis, iritis, inflammatory bowel syndrome, sacroiliitis, metabolic syndrome or positive test for human leukocyte antigen (HLA) B 27.
6. Any condition that, in the investigator's opinion would impact participant safety and/or a participant's ability to complete all study related procedures. (e.g., psychiatric illness, drug addiction, alcoholism, etc.)
7. Infection with hepatitis B or C, human immunodeficiency virus (HIV), human T-lymphotropic virus (HTLV) or syphilis
8. Participants diagnosed with cancer with or without chemotherapy treatment
9. Women who are pregnant or nursing
10. Ongoing or recent (within the previous 6 months) participation in a clinical research study.
11. Participants diagnosed having uncontrolled systemic diseases
12. Use of any medications not permitted in the study (see Excluded Medications)
13. Participants currently using other active treatments for tendinosis other than physiotherapy (e.g., acupuncture, trigger point therapy, chiropractic treatments, glyceryl trinitrate patches) during study or within 3 months prior to Visit 1
14. Unresolved litigation or insurance claims (e.g., Workers Compensation, WorkSafe BC, etc.) involving the Achilles tendinopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-05; Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 6 months post-injection
  Comparison of the safety profile between RCT-01/placebo treatment groups. The safety profile is defined by the incidence, relationship to treatment, severity and seriousness of adverse events.

SECONDARY OUTCOMES:
Victorian Institute of Sport Assessment - Achilles (VISA-A) questionnaire | 6 months post-injection
Visual analog scale (VAS) | 6 months post-injection
  pain on palpation and pain on loading (running/jumping)
Modified Tegner Activity Scale | 6 months post-injection
SF-36 questionnaire | 6 months post-injection
  quality of life questionnaire
Tendon condition (appearance, biomechanics, and blood flow) | 6 months post-injection
  Ultrasound imaging will be utilized to measure: echogenicity, hyperemia or neovascularisation, anechoic regions/intratendinous tears, intratendinous calcification, any irregularities to the cortical bone at insertion, and tendon thickness

CONTACTS AND LOCATIONS:
Overall Officials: D R Lloyd-Smith, MDCM, Principal Investigator — University of British Columbia
Locations (1):
- Allan McGavin Sports Medicine Centre, Vancouver, British Columbia, Canada

REFERENCES:
- See also: RepliCel Life Sciences, Inc. Website — http://www.replicel.com
- See also: Study information site for potential participants — http://www.tendonstudy.com